CLINICAL TRIAL: NCT06063278
Title: Step by Step Group Therapy for Bulimia Nervosa: Effectiveness and Mechanisms of Change.
Acronym: SBSBN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-BUL-2021-144
Record Dates: First submitted 2022-04-28; First posted 2023-10-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-11

CONDITIONS: Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BN Group (Experimental): Patients will take part of a Therapeutic BN Group
  Interventions: Behavioral: l Group Therapy for BN.
- Waiting List (No Intervention): Participants will be in the waiting list.

INTERVENTIONS:
Behavioral: l Group Therapy for BN. — 9 to 10 group sessions of 90 to 120min each
  Arms: BN Group

SUMMARY:
This a pseudo-randomized clinical trial that examines if a specific group therapy for BN is effective in improving its symptomatology, and what variables mediate such improvements. To do so a sample of 100 patients with BN will be pseudorandomized in a Group Therapy for BN or in a control waiting list group. Patients will be assessed at baseline, at the end of the group therapy and at 2 year follow up.

DETAILED DESCRIPTION:
This is a controlled non randomized study that will compare a group of patients with BN that participate in the SBS group therapy with a group of BN patients who will be in wait list as a control condition.

Patients for this single center trial will be recruited from the outpatient facility of the Hospital de la Santa Creu I Sant Pau (Barcelona, Spain).

After assessed for eligibility participants will be given a set of self -report questionnaires. After the questionnaires are completed participants will be allocated to wait list condition or to the treatment arm. Time between assessment and starting the SBS group will be a month or least. Participants will be administered the same questionnaires the following month after finishing the treatment or after 3 to 4 months after the first assessment for the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Bulimia Nervosa

Exclusion Criteria:

* Not understanding Spanish or Catalan Language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Eating Attitudes Test, E-40. | 3 months
  A self report questionarie that assesses eating disorder symptomatology. The range of scores is 0-78. Higher scores mean higher eating disorders sympthoms.
Eating Disorder Inventory, EDI | 3 months
  A self report questionarie that assesses eating disorder symptomatology. The range of scores is 0-192. Higher scores mean higher eating disorders sympthoms
Bulimic Investigatory Test Edinburgh, BITE | 3 months
  A self report questionarie that assesses bulimia nervosa symptomatology.The range of scores is 0-30. Higher scores mean higher bulimic sympthoms
Body Shape Questionnaire, BSQ-34 | 3 months
  A self report questionarie that assesses eating disorder symptomatology. The score is ranging between 34-204 points. Higher scores point to an increased level of concern on body shape.

SECONDARY OUTCOMES:
Working alliance Inventory -short, WAIS. | 3 months
  A self report questionarie that assesses bulimia nervosa symptomatology. Values range from 12 to 84. Hihger scores meaning higher therapeutic alliance.
Autism-Spectrum Quotient, AQ | 3 months
  A self report questionarie that assesses autistic traits. The range of scores is 0 to 50. Higher scores mean higher autistic traits.
Quality of Life Enjoyment and Satisfaction Questionnaire, Q-LES-Q. | 3 months
  A self report questionarie that assesses quality of life. The range of scores is 0-100. Higher scores mean higher quality of life.
Beck Depression Inventory, BDI-II | 3 months
  A self report questionarie that assesses depressive symptoatology. The range of scores is 0-83. Higher scores mean higher depressive symptoms.
Rosenberg Self-Esteem Scale, RSE. | 3 months
  A self report questionarie that assesses self steem. The scale ranges from 0-30. Higher scores mean higher self-esteem. The range scores is 0-60.
State -Trait Anxiety Inventory, STAI. | 3 months
  A self report questionarie that assesses anxiety. Higher scores mean higher anxiety.
Difficulties in Emotion Regulation Scale (DERS). | 3 months
  A self report questionarie that assesses emotion regulation difficulties. The scale ranges from 28-40. H igher scores indicate more difficulty in emotion regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agh T, Kovacs G, Supina D, Pawaskar M, Herman BK, Voko Z, Sheehan DV. A systematic review of the health-related quality of life and economic burdens of anorexia nervosa, bulimia nervosa, and binge eating disorder. Eat Weight Disord. 2016 Sep;21(3):353-364. doi: 10.1007/s40519-016-0264-x. Epub 2016 Mar 4. PMID 26942768
- [Background] - Andrade-González, N., & Fernández-Liria, A. (2016). Spanish adaptation of the working alliance inventory-short (WAI-S). Current Psychology, 35(1), 169-177.
- [Background] Fairburn CG, Bailey-Straebler S, Basden S, Doll HA, Jones R, Murphy R, O'Connor ME, Cooper Z. A transdiagnostic comparison of enhanced cognitive behaviour therapy (CBT-E) and interpersonal psychotherapy in the treatment of eating disorders. Behav Res Ther. 2015 Jul;70:64-71. doi: 10.1016/j.brat.2015.04.010. Epub 2015 Apr 22. PMID 26000757
- [Background] Hay P. A systematic review of evidence for psychological treatments in eating disorders: 2005-2012. Int J Eat Disord. 2013 Jul;46(5):462-9. doi: 10.1002/eat.22103. PMID 23658093
- [Background] Polnay A, James VA, Hodges L, Murray GD, Munro C, Lawrie SM. Group therapy for people with bulimia nervosa: systematic review and meta-analysis. Psychol Med. 2014 Aug;44(11):2241-54. doi: 10.1017/S0033291713002791. Epub 2013 Nov 15. PMID 24238470